CLINICAL TRIAL: NCT04503473
Title: Locomotor Recovery Following Traumatic Brain Injury
Acronym: TBI_IU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, George Hornby, Professor of Physical Medicine & Rehabilitation, Indiana University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1911962819
Record Dates: First submitted 2019-12-16; First posted 2020-08-07 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Traumatic Brain Injury (TBI)
Keywords: Traumatic Brain Injury; TBI; Walking
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Intervention Model Description: Baseline characteristics and training parameters (steps, intensity parameters) will be compared between treatment groups using independent group comparisons. (ANOVA, Kruskal-Wallis, or Chi-squared tests as appropriate).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Intensity Stepping Training (Experimental): The primary goal will be to perform continuous stepping while maintaining HR within 70-85% maximum predicted HR (if patients are deconditioned, PTs will gradually increase intensity to desired levels as tolerated). We will also record Ratings of Perceived Exertion (RPE) every 3-5 minutes, with goals of 15-18. Sessions will be divided into ~10 minute increments (~25% of sessions) between speed-dependent treadmill training (described above for treadmill stepping), skill-dependent treadmill training, overground training, and stair climbing.
  Interventions: Behavioral: High Intensity Stepping Training
- Conventional Therapy (Active Comparator): Participants provided conventional therapy will perform various standardized exercise tasks during 40 minutes of 1 hr sessions. The type of therapeutic activities is based on published normative data of typical activities performed during clinical physical therapy sessions with focus on strengthening activities (25% of session); balance activities (25%); locomotor activities (25%), and combined stretching exercises (10-15%) and transfers (10-15%). Intensity of activities will be targeted at 30-40% of their HR reserve in attempts to maintain consistent intensities between training groups.
  Interventions: Behavioral: Conventional Therapy

INTERVENTIONS:
Behavioral: High Intensity Stepping Training — The goals will be to maximize stepping activity at high intensities for 40 minutes per 1 hour session, with rest breaks as needed
  Conventional Therapy: : Participants provided conventional therapy will perform various standardized exercise tasks during 40 minutes of 1 hr sessions
  Other Names: HIT
  Arms: High Intensity Stepping Training
Behavioral: Conventional Therapy — Participants provided conventional therapy will perform various standardized exercise tasks during 40 minutes of 1 hr sessions
  Arms: Conventional Therapy

SUMMARY:
The purpose of this study is to investigate the effectiveness of two different walking training interventions on the recovery of strength, mobility, walking and other measures of health in individuals following traumatic brain injury. During this study, participants will aim to complete up to 15 training sessions over 4-5 weeks of each intervention with at least a 4 week break between interventions. Each training session will last approximately 1 hour, while testing sessions performed at the beginning and end of each intervention will last approximately 3-4 hours. Participation in this research study may last up to 6 months including screening and baseline testing. The possible benefits to participant from participation in this study include increased strength of the participants leg muscles and improved walking ability

DETAILED DESCRIPTION:
The primary goal of the proposed study is to identify the contributions of the amount of task-specific practice on locomotor (i.e., walking) recovery in patients with (> 6 Months) traumatic brain injury (TBI). The investigator will do this by building on our previous work directed towards identifying the essential exercise training parameters that maximize locomotor recovery. Consistent with principles of motor learning and exercise physiology, the investigator contend that certain training (i.e., dosage) parameters of physical rehabilitation, including the type (specificity) and amount of task practice, are critical to mobility outcomes following neurological injury. Previous work suggests these training parameters may influence locomotor recovery in patients with other neurological disorders (i.e., stroke), although few studies have attempted to delineate similar contributions of amount of task-specific practice in neurologic injury. Indeed, no studies have carefully controlled these training parameters during physical rehabilitation of patients with neurologic injury, and such interventions are rarely utilized in the clinical setting. Reasons for these knowledge gaps from other rehabilitation studies to patients with neurologic injury or lack of clinical implementation are unclear, but may be due to adherence to traditional rehabilitation theories. One concern is that practicing only stepping tasks reduces attention towards hallmark physical impairments following neurologic injury, such as loss of strength or postural stability, which are considered primary determinants of decreased mobility. Only a few studies have addressed whether providing only structured stepping training can mitigate these impairments without their explicit practice, but not in the neurologic injury population. A related concern is that focused stepping training without significant attention towards impairments or gait quality may exaggerate altered movement strategies, which could be reinforced with repeated practice. However, there is little data to suggest "worsening" of abnormal gait patterns following high intensity training. Rather, recent findings suggest patients demonstrate more normal kinematics. If focused task specific (i.e., stepping) training is to be applied clinically, participant must delineate its contributions towards improving locomotor function, and their effects on underlying impairments and gait kinematics.

Central hypotheses are that stepping training in TBI results in:1) greater locomotor gains as compared to non-specific interventions; 2) gains in selected impairments underlying gait dysfunction (i.e., strength and metabolic capacity and efficiency); and, 3) improvements in gait quality. To test these hypotheses, the proposed crossover, assessor-blinded, randomized clinical trial (RCT) is designed to test the effects of specificity of rehabilitation training applied early-post-stroke. In this RCT, patients > 6 post-TBI will be allocated ≤ 15 sessions over approximately 4-5 weeks of high-intensity stepping training or conventional therapy. Importantly, training intensity will be held constant to account for this potential confounding factor. Blinded assessments will be performed prior to and following each training paradigm.

ELIGIBILITY:
Inclusion Criteria:

* > 6 months post traumatic brain injury
* 18-75 years old
* ability to walk without physical assistance
* Self selected walking speed of 0.01-1.0 m/s

Exclusion Criteria:

* <18 years old
* >75 years old
* self selected walking speed of > 1.0 m/s
* < 3 months from botulinum toxin injection
* Above the knee brace
* Currently receiving physical therapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Gait speed | Baseline 1, Post 6 weeks, Baseline 2, Post 6 weeks
  Gait speed is valid, reliable, and sensitive measures related to overall functional ability, and will be assessed by blinded rates. This measure will be performed by blinded assessors who do not participate in the training. Gait speed will be measured at self-selected speeds (SSS; instructions to "walk at normal comfortable pace") and fastest-possible speed (FS: "as fast as you safely can") using the Zeno Walkway (Protokinetics, Haverton, PA).
Change in Endurance | Baseline 1, Post 6 weeks, Baseline 2, Post 6 weeks
  Endurance is valid, reliable, and sensitive measures related to overall functional ability, and will be assessed by blinded rates. This measure will be performed by blinded assessors who do not participate in the training. Gait endurance will be tested using the 6MWT (m) with instructions similar to SSS to minimize fall risk.

SECONDARY OUTCOMES:
Change in Strength | Baseline 1, Post 1 after 6 weeks, Baseline 2, Post 6 weeks
  • Peak volitional strength - We will assess strength while subjects are seated in an adjustable height chair of a testing apparatus. Three trials of peak isometric volitional hip, knee and ankle torques will be determined bilaterally with significant verbal encouragement for 3-5 sec, and > 1 min duration between trials.
Change in gait quality | Baseline 1, Post 6 weeks, Baseline 2, Post 6 weeks
  Gait kinematics: Lower limb kinematics will be collected using an 8-camera motion capture system and 3-dimensional movement of 1" reflective markers affixed to the pelvis/legs. Spatiotemporal metrics will be extracted from the data, with primary measures of peak speed, stride length, cadence. All measures will be compared between fastest speeds achieved at BSL and POST, and at POST speeds matched to BSL peak speed to allow kinematic comparisons while controlling for speeds.
Change in metabolic capacity | Baseline 1, Post 6 weeks, Baseline 2, Post 6 weeks
  peak metabolic capacity will be observed during graded exercise testing on a treadmill wtih peak oxygen consumption

CONTACTS AND LOCATIONS:
Overall Officials: George Hornby, PhD, Principal Investigator — Indiana University
Locations (1):
- Rehabilitation Hospital of Indiana, Indianapolis, Indiana, United States

REFERENCES:
- [Derived] Plawecki A, Henderson CE, Lotter JK, Shoger LH, Inks E, Scofield M, Voigtmann CJ, Katta-Charles S, Hornby TG. Comparative Efficacy of High-Intensity Training Versus Conventional Training in Individuals With Chronic Traumatic Brain Injury: A Pilot Randomized Controlled Study. J Neurotrauma. 2024 Apr;41(7-8):807-817. doi: 10.1089/neu.2023.0494. Epub 2024 Jan 25. PMID 38204184